CLINICAL TRIAL: NCT05551364
Title: Usabilidad y Efectividad Del Exoesqueleto ATLAS2030 en Variables físicas, Emocionales y Funcionales en niños Con parálisis Cerebral
Brief Title: Usability and Effectiveness of the ATLAS2030 Exoskeleton in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Collaborators: Hospital Miguel Servet (Other); ATADES (Unknown); Universidad de Zaragoza (Other); Spanish National Research Council (Other Government); Fundación Bobath Madrid (Unknown); ATENPACE Madrid (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A30-ATADES-CP
Record Dates: First submitted 2022-09-02; First posted 2022-09-22 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Palsy
Keywords: exoskeleton; paediatric; gait; robotic gait assited training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment (No Intervention): The children will continue with their current rehabilitation program
- Treatment with the ATLAS 2030 Exoskeleton (Experimental): The children will receive 2 hours of exoskeleton ATLAS 2030 gait training a week for 3 months
  Interventions: Device: ATLAS 2030 exoskeleton

INTERVENTIONS:
Device: ATLAS 2030 exoskeleton — Individualized Rehabilitation Treatment with the ATLAS 2030 Exoskeleton consists of the following phases:
  1. Telephone contact phase (1 session)
  2. Inclusion Phase (1 session)
  3. Signing of informed consent (1 session)
  4. Initial Evaluation Phase (1 session)
  5. Treatment Phase (1st part) (7 sessions)
  6. Monthly Evaluation Phase (1 session)
  7. Treatment Phase (2nd part) (7 sessions)
  8. Monthly Evaluation Phase (1 session)
  9. Treatment Phase (3rd part) (7 sessions)
  10. Final Evaluation Phase and results (2 sessions)
  Arms: Treatment with the ATLAS 2030 Exoskeleton

SUMMARY:
The main objective of this study is to assess the usability and efficacy of receiving therapy with the peaditric exoskeleton ATLAS 2030in children with gait impairment due to a cerebral palsy condition. It will be valued the impact of rehabilitation with the exoskeleton at the physical level on parameters such as joint range, spasticity, as well as the impact in quality of life. It is also assessed the impact at the level of functionality of the participants, through the administration of different functional assessment scales.

ELIGIBILITY:
Inclusion Criteria:

* Medical authorization to for standing, gait training and weight bearing.
* Maximum user weight of 35 kg.
* Length of the thigh (distance from the greater trochanter to the lateral condyle of the tibia) from 24cm to 33cm.
* Tibia leg length (distance from the lateral condyle of the tibia to the lateral malleolus) from 23cm to 32cm.
* Hip width (between greater trochanteres) less than or equal to 35 cm.
* Do not have an allergy to any of the ATLAS materials: cotton, nylon, polyester, polyamide, polyethylene or propylene.
* Ability to achieve the neutral position of the ankle, during the use of the device with or without technical aids.
* Informed consent signed by legal guardians.
* Confirmed diagnosis of cerebral palsy affecting the ability to walk.
* Stable medical condition without modifications of the specific medication for the disease in the last 6 months, and other additional medication in the last month.
* Patient in follow-up according to the normal standards recommended for his illness.

Exclusion Criteria:

* More than 20º of hip flessum at the time of using the exoskeleton.
* More than 20º of knee flessum at the time of using the exoskeleton.
* Severe skin lesion on parts of the lower extremities that are in contact with the device.
* Scheduled surgery (rachis, limbs) for the duration of the study or surgery performed (rachis, extremities) in the last 6 months.
* History of fracture without trauma. History of bone fracture traumatic in lower extremities or pelvic girdle in the last 3 months.
* Refusal of the patient or legal guardian to include the child in the study.
* Skin problems (diseases, allergies, sensitivity ...) that prevent the use of exoskeleton accessories on the patient's skin.
* Spasticity equal to 4 on the Modified Ashworth Scale at the time of use of the device.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Classification System | Every month up to 3 months
  To indentify the diffrent levels of the Gross Motor Function Classification System who can use the ATLAS 2030 exoskeleton. The Gross Motor Function Classification System goes from Level 1 (can walk indoors and outdoors and climb stairs without using hands for support; can perform usual activities such as running and jumping; has decreased speed, balance and coordination) to Level 5 (has physical impairments that restrict voluntary control of movement and the ability to maintain head and neck position against gravity; is impaired in all areas of motor function; cannot sit or stand independently, even with adaptive equipment; cannot independently walk, though may be able to use powered mobility)
To quantify number of steps taken within the device | Every session up to 28 sessions
  Quantity of steps taken within the exoskeleton
Changes in joint range of motion | Every session up to 28 sessions
  To evaluate the joint range of motion changes at the hip, knee and ankle after the ATLAS 2030 use measured by goniometer
Changes in spasticity | Every session up to 28 sessions
  To evaluate spasticity changes at the lower limb muscle groups after ATLAS 2030 use by Modified Asworth Scale
Changes in the Six-Minute Walking Test performance | Every month up to three months
  To assess changes in the distance the child can walk in six minutes by using the Six-Minute Walking Test
Changes in the 10 Meters Walking Test performance | Every month up to three months
  To assess changes in the time needed to walk 10 meters by using the 10 Meters Walking Test
Changes in the time walked within the device | Three months
  To assess possible changes in the time walked within the device
Changes in the Gross Motor Function Measure 88 for children with cerebral palsy (GMFM-88) | Every month up to three months
  To evaluate possible changes in the gross motor function after 3 months of ATLAS 2030 use twice a week where a higher score means child´s gross motor function is better
Changes in the Functional Independence Measure for Children (WeeFim) | Every month up to three months
  To evaluate possible changes in the overall functionality after 3 months of ATLAS 2030 use twice a week by using the Functional Independence Measure for Children where a higher score means the child is more functional, more independant
Cerebral Palsy Quality of Life | Three months
  To assess possible changes in the quality of life of the children after using the ATLAS 2030 for 3 months twice a week by using the Cerebral Palsy Quallity of Life scale where a higher percentage means a better quality of life

SECONDARY OUTCOMES:
Safety of the ATLAS 2030 | at study completion
  Measured as the occurrence of adverse events such as onset of pain, fatigue, presence of falls or alteration of the integrity of the user's skin, by the use of the device.
The Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) | at study completion
  To assess both professionals and patients´satisfaction when using the ATLAS 2030
Acceptability | at study completion
  Measured through the dropout rate of the participants.
Accessibility | at study completion
  Measure such as the relationship between the number of patients recruited and potential patients who were not recruited

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Colegio de Educación Especial San Martín de Porres (ATADES), Zaragoza, Aragon
  - ATENPACE, Madrid
  - Centre for Automation and Robotics, Marsi Care, Madrid
  - Fundación Bobath, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
  - Universidad de Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No